CLINICAL TRIAL: NCT03854682
Title: Surgical or Non-surgical Treatment of Plantar Fasciitis - A Randomized Clinical Trial
Brief Title: Surgical or Non-surgical Treatment of Plantar Fasciitis
Acronym: SOFT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Carsten Jensen, Associate professor, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 67030
Record Dates: First submitted 2019-02-08; First posted 2019-02-26 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Fasciitis, Plantar, Chronic
MeSH Terms: conditions — Fasciitis, Plantar | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: A prospective, blinded, parallel-group trial with balanced randomization [1:1], in accordance with CONSORT
Who Masked: Investigator, Outcomes Assessor
Masking Description: Blinding to treatment allocation of patients, physiotherapists (health care providers) will not be possible due to the nature of the interventions. However, independent data collectors will be responsible for baseline and follow-up assessments, while all self-reported outcome measures will be made available to the patients electronically, and responses entered into a database identified by identification numbers only. The data analyst will be unaware of the treatment allocation as data will be analyzed using recoded identification numbers. The recoding will be performed by an independent person.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgical (Experimental): Radiofrequency microtenotomy (RF): A longitudinal incision of about 3 cm will be made over the most tender part of the foot taking care to avoid the weight bearing part of the sole, and the tissues dissected down to the affected plantar fascia. After initiating sterile isotonic saline flow of 1 drop every 1-2 s from a line connected to the RF system, the TOPAZ tip will be placed onto the fascia and the micro debridements carried out in a grid like pattern on and throughout the symptomatic fascia area. After debridement, the wound will be irrigated with copious amounts of normal saline solution and closed in layers. A local anaesthetic will be injected into the skin and subcutaneous tissues around the wound and standard wound dressings will be applied
  Interventions: Procedure: Radiofrequency microtenotomy
- Non-surgical (Active Comparator): Strength training: Consists of one-legged heel lift to primarily activate the windlass effect and increase the mechanical stress on the tendon. The exercise is performed on a step, a thick book or the like, so the heel movement finishes below the horizontal level. The exercise is performed every other day with as many sets as possible and as heavy as possible, but not heavier than eight repetitions can be performed per. set. The load progressed from two to one leg +/- backpack. The exercise is performed as 3 s/2 s / 3 s concentric, isometric and eccentric respectively followed by 2 min rest. Patients continue to exercise 4 weeks after patient acceptable symptom state (PASS) has been achieved
  Interventions: Behavioral: Strength training

INTERVENTIONS:
Procedure: Radiofrequency microtenotomy — A longitudinal incision of about 3 cm will be made over the most tender part of the foot taking care to avoid the weight bearing part of the sole, and the tissues dissected down to the affected plantar fascia. After initiating sterile isotonic saline flow of 1 drop every 1-2 s from a line connected to the RF system, the TOPAZ tip will be placed onto the fascia and the micro debridements carried out in a grid like pattern on and throughout the symptomatic fascia area. After debridement, the wound will be irrigated with copious amounts of normal saline solution and closed in layers. A local anaesthetic will be injected into the skin and subcutaneous tissues around the wound and standard wound dressings will be applied
  Arms: Surgical
Behavioral: Strength training — Non-surgical treatment consists of one-legged heel lift to primarily activate the windlass effect and increase the mechanical stress on the tendon. The exercise is performed on a step, a thick book or the like, so the heel movement finishes below the horizontal level. The exercise is performed every other day with as many sets as possible and as heavy as possible, but not heavier than eight repetitions can be performed per. set. The load progressed from two to one leg +/- backpack. The exercise is performed as 3 s/2 s / 3 s concentric, isometric and eccentric respectively followed by 2 min rest. Patients continue to exercise 4 weeks after patient acceptable symptom state (PASS) has been achieved
  Other Names: Resistance training
  Arms: Non-surgical

SUMMARY:
Plantar fasciitis (PF) is one of the most common causes of heel pain in 40-60 year old people. Approximately 10% of the population is affected by the disorder and the PF prevalence is 3.6-7.0%. The risk factors include decreased ankle dorsiflexion, overweight (BMI> 27), pronated foot position, and prolonged work and activity-related weight bearing. The condition affects both active and less active people.

The typical symptoms are pain around the attachment of the foot's tendon mirror (fascia plantaris), especially the medial part. The pain is well defined and occurs during weight bearing activities or during the first steps after rest. The walking pattern is changed to relieve pain. Ultrasound scan is used to confirm the diagnosis (thickened tendon mirror> 4 mm). The condition is described as inflammatory, but the relationship between the initial inflammatory condition and the chronic tendon mirror overload injury (fasciopathy) is unknown and marked by degenerative changes.

Although the majority of people improve within 1-2 years, the long-term prognosis is unknown. People with symptoms lasting > 7 months have poor prognosis and should be offered other treatment. Non-surgical treatment is often first line of treatment followed by surgical treatment.

In this clinical trial investigators compare pain levels (FHSQ-DK) in people, who receive surgical treatment (radiofrequency microtenotomy, shoe inserts and patient education) and people who receive non-surgical treatment (strength training, shoe inserts and patient education) with a primary end-point at 6 months. The hypothesis is that surgical treatment is better than non-surgical treatment measured by FHSQ-DK (pain)

DETAILED DESCRIPTION:
To be completed later

ELIGIBILITY:
Inclusion Criteria:

* VAS pain score > 30 within last 7 days
* Plantar heel pain> 7 months
* Palpation soreness fascia plantaris at heel
* Plantar heel pain during first steps (First-step sign)
* Read and understand Danish

Exclusion Criteria:

* Systemic diseases or neuropathy
* Diabetes
* Pregnant
* Previous heel surgery on same foot
* Cortisone injections within past 3 months
* Bilateral symptom onset within past 7 days
* Signs of tarsal tunnel
* Facia plantaris thickness of less than 4 mm
* Performed message / head recovery / stretching within the past month
* Any treatment for plantar pain within the past 3 months
* Other reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in the Foot Health Status Questionnaire (FHSQ) | Change from baseline at 6 months
  Subdomain foot pain score range 0-100, low values represent worse conditions

SECONDARY OUTCOMES:
The Foot Health Status Questionnaire (FHSQ) | Change from baseline at 6 months
  Subdomains (foot related function, footwear and general foot health perception). Subdomain scores range from 0-100, low scores represent worse conditions
Visual Analog Scale (VAS) | Change from baseline at 6 months
  Pain and scores range from 0-100, low values represent worse conditions
Global Percieved Effect (GPE) | 1,3,6,12 months post-intervention
  A questionnaire using a 7-point likert scale to asses change in symptoms. The scores are categorized into (1-2 = deterioration of symptoms, 3-5 = Neutral, 6-7 improvement of symptoms).
Physical Activity Questionnaire (IPAQ) | Change from baseline at 6 months
  Participation in sports and activities of daily living measured as MET-minutes/day or MET-minutes/week. Low MET-scores indicate limited activity. MET = metabolic equivalent of task

OTHER OUTCOMES:
Compliance with the prescribed intervention | 6 months
  Tracking adherence to exercise and reasons for non-complience
Complications and side-effects | 6 months
  Review of medical records for complications and side-effects

CONTACTS AND LOCATIONS:
Locations (1):
- Lillebaelt Hospital, Kolding, Kolding, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moller S, Riel H, Wester J, Simony A, Viberg B, Jensen C. Surgical or non-surgical treatment of plantar fasciopathy (SOFT): study protocol for a randomized controlled trial. Trials. 2022 Oct 4;23(1):845. doi: 10.1186/s13063-022-06785-w. PMID 36195936